CLINICAL TRIAL: NCT06410365
Title: Impact of Intrathecal Versus Intravenous Dexmedetomidine Adjuvant to Bupivacaine in Elective Cesarian Section
Brief Title: Impact of Intrathecal vs Intravenous Dexmedetomidine
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Muhammad Ilyas (Other)
Responsible Party: Sponsor-Investigator, Muhammad Ilyas, Assistant professor, Watim Medical & Dental College
Organization: Watim Medical & Dental College (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: WM&DCR/R&D(ERB)/2023/64
Record Dates: First submitted 2024-04-29; First posted 2024-05-13 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Nausea and Vomiting, Postoperative
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Dexmedetomidine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intrathecal dexmedetomidine+ bupivacaine (Experimental): intrathecal bupivacaine 0.75%(1.2ml+plus 5 μg Dex (diluted in N/S up to the volume of 1 ml intrathecally once
  Interventions: Drug: Dexmedetomidine injection
- intravenous dexmedetomidine+ bupivacane (Experimental): intravenous dexmedetomidine 1mcg/kg in normal saline + intrathecal .75% bupivacaine (1.2ml)
  Interventions: Drug: Dexmedetomidine injection

INTERVENTIONS:
Drug: Dexmedetomidine injection — Comparison of intravenous and intrathecal route of dexmedetomidine
  Other Names: Bupivacaine

SUMMARY:
The purpose of this research is to evaluate the impact of intrathecal dexmedetomidine in comparison with intravenous route in patients undergoing cesarean section.

Alternate hypothesis :Dexmedetomidine is more effective when given intrathecally as adjuvant to bupivacaine in elective cesarean section Null Hypothesis: Dexmedetomidine is more effective when given intravenously as adjuvant to bupivacaine in elective cesarean section Study Design: Randomized controlled trial Study setting: Watim General Hospital Study Duration: 18 months after synopsis approval Sampling technique: Simple random sampling Sample Size: Using the Open Epi program, a sample size of 60 patients (30 in each group) was determined with a 95% confidence interval and 80% power.

Inclusion Criteria:

* Pregnant women between ages 18-35 years
* Belongs to ASA class I or II
* Subjected to elective C-section

Exclusion Criteria:

* Any history of gastrointestinal disease diabetes, thyroid disease, hypertension, obesity, or anemia
* History of alcohol or drug abuse;
* Major complications of pregnancy
* Patients have contraindication to spinal block or allergic to any of drug

DETAILED DESCRIPTION:
Introduction Cesarean section under spinal anesthesia has gained worldwide popularity in the past two, three decades as it provides quick, intense and balanced anesthesia. Patients may avoid the dangers of general anesthesia by having a cesarean section while still receiving anesthetic and pain relief via spinal anesthesia Patients still experience problems during surgical operations due to adverse effects produced by spinal anesthesia, such as nausea, vomiting and shivering, even though the risk is lower than that of general anesthetic One research estimates that as many as 55 percent of people shiver at some point throughout their lives .There may be adverse consequences on heart rate, oxygen saturation, and blood pressure from excessive shivering. Cardiopulmonary insufficiency increases the risk for potentially fatal side effects While there has been much research on nausea and vomiting after epidural anesthesia, less attention has been paid to IONV during the procedure itself Patients' comfort is diminished, hospital stays are prolonged, and more expenses are incurred when nausea and vomiting occur during surgery and remain thereafter. Considerable attention should be paid to this issue because of the seriousness of its potential outcomes, which include, among others, dehydration, electrolyte imbalance, wound dehiscence, venous hypertension and bleeding, esophageal rupture, airway obstruction, and aspiration pneumonia. In several types of surgeries, patients often have nausea and vomiting afterward However, caesarean sections performed with regional anesthesia have this issue more often . There are several factors that might put a patient at risk for IONV, including increased intragastric pressure, hypotension, extending the peritoneum (exteriorization of the uterus), extensive surgical manipulation and visceral stimulation, the use of opioids, the use of uterotonic drugs, and the patient's mental health. The hypotension that occurs during spinal, epidural, or spinal-epidural (combined) anesthesia is a major risk factor for ischemic optic neuropathy of the visual system. Procedure-specific factors that may lead to IONV include peritonealization, exteriorizing the uterus for suturing, and peritoneal cleaning IONV has an estimated 80 percent prevalence. As a result, preventative medicine is essential . Treatment rather than prevention has been the primary focus of previous IONV research. It seems that IONV may be improved by using a combination of preoperative and intraoperative midazolam and propofol, closely monitoring hypotension, attaining a good anesthetic block, doing surgery gently, and using uterotonic drugs sparingly.

Postoperative pain is still a major problem in healthcare all around the world, despite developments in anesthesiology and surgical methods. Poor pain management after surgery is linked to several unfavorable results, including patient dissatisfaction, low quality of life, slowed healing, and increasing reliance on drugs . Intrathecal block is the most popular method for anesthetizing patients undergoing C-sections, which is the most frequent surgical operation for women of childbearing age. Increased protection for both mother and child, a strong motor and sensory block, a low failure rate, and a reasonable price tag are just a few of the benefits it provides. Subarachnoid block, when done just with local anesthetics, has the fundamental drawback of providing only temporary relief from postoperative pain due to its limited duration of action. Adjuvants are often used to enhance the duration of analgesia by enhancing the quality of the block and lengthening the duration of analgesia . Intrathecally administering dexmedetomidine, a highly selective alpha-2 agonist, in combination with hyperbaric bupivacaine results in a much longer duration of analgesia and an improved safety profile .Studies on full-term patients having spinal anesthesia for elective caesarean sections indicated that the combination of Dexmedetomidine and bupivacaine was just as effective as morphine and bupivacaine for maintaining pain relief for a longer period of time showed that among ASA I or II patients undergoing caesarean delivery, the duration of analgesia produced by bupivacaine + Dexmedetomidine was significantly longer than the length provided by bupivacaine + placebo. Dexmedetomidine patients also had considerably decreased postoperative rescued sufentanil intake compared to those in the control group.

We expect that the addition of dexmedetomidine as an adjuvant to intrathecal hyperbaric bupivacaine would enhance intraoperative blockade conditions during cesarean section, extend postoperative sensory block, reduce nausea vomiting and shivering without affecting the motor block and with minimal additional adverse effects.

Data Collection:

Participant's demographic and clinical information will be obtained through a questionnaire and the patient will be randomly divided into two groups using lottery method. Participants in Group A will receive an intravenous dose of dexmedetomidine diluted in 20 milliliters of saline, with 1 milliliter withdrawn from a 2-milliliter syringe. Group B will receive intravenously one milliliter of 0.9% isotonic saline in a two milliliter syringe. The participant will be given a subarachnoid block in accordance with standard operating procedure. Group A will receive intrathecal 0.75% bupivacaine (1.2ml +1 ml N/S) and group B will receive intrathecal bupivacaine 0.75%(1.2ml+plus 5 μg Dex (diluted in N/S up to the volume of 1 ml intrathecally. T4-5 block will be achieved by turning the patient supine with left uterine displacement. . Intraoperative nausea and vomiting will be assessed using a a 4-point scale (0 = absent; 1 = mild; 2 = moderate; 3 = severe) Postoperative pain will measured using a numeric pain rating scale (0=no pain, 1-3=mild pain, 4-6=moderate pain, and 7-10=severe pain) every 30 minutes in the postoperative care unit until the patient demanded their first analgesic dose, which will serve as the study's cut-off point. Injectable Ketorolac 30 mg will be used as a rescue analgesic

Data Analysis:

SPSS-23 will be used for the statistical analysis of the data. The duration of post-operative analgesia will be compared between the two groups using an independent sample t-test. Using stratification, we will be able to regulate potential confounding variables. To compare how long patients needed pain relief after surgery among groups, an independent samples t-test will be used after stratification. The cutoff for significance will be set at P≤0.05.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between ages 18-35 years
* Belongs to ASA class I or II
* Subjected to elective C-section

Exclusion Criteria:

* Any history of gastrointestinal disease diabetes, thyroid disease, hypertension, obesity, or anaemia
* History of alcohol or drug abuse;
* Major complications of pregnancy
* Patients have contraindication to spinal block or allergic to any of drug

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the impact of clinical efficacy of intrathecal versus intravenous dexmedetomidine on intraoperative nausea vomiting,shivering and postoperative pain | during cesarean section surgery
  Intraoperative nausea and vomiting will be assessed using a a 4-point scale (0 = absent; 1 = mild; 2 = moderate; 3 = severe) Postoperative pain will measured using a numeric pain rating scale (0=no pain, 1-3=mild pain, 4-6=moderate pain, and 7-10=severe pain) every 30 minutes in the postoperative care

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 6 months after completion of study

REFERENCES:
- [Background] Semiz A, Akpak YK, Yilanlioglu NC, Babacan A, Gonen G, Cam Gonen C, Asiliskender M, Karakucuk S. Prediction of intraoperative nausea and vomiting in caesarean delivery under regional anaesthesia. J Int Med Res. 2017 Feb;45(1):332-339. doi: 10.1177/0300060516680547. Epub 2017 Jan 17. PMID 28222642
- [Background] Harris PH. General versus spinal anaesthesia. Br Med J (Clin Res Ed). 1985 Apr 27;290(6477):1286. doi: 10.1136/bmj.290.6477.1286-a. No abstract available. PMID 3921186
- [Background] Miao S, Shi M, Zou L, Wang G. Effect of intrathecal dexmedetomidine on preventing shivering in cesarean section after spinal anesthesia: a meta-analysis and trial sequential analysis. Drug Des Devel Ther. 2018 Nov 2;12:3775-3783. doi: 10.2147/DDDT.S178665. eCollection 2018. PMID 30464408
- [Background] Bi YH, Wu JM, Zhang YZ, Zhang RQ. Effect of Different Doses of Intrathecal Dexmedetomidine as an Adjuvant Combined With Hyperbaric Ropivacaine in Patients Undergoing Cesarean Section. Front Pharmacol. 2020 Mar 20;11:342. doi: 10.3389/fphar.2020.00342. eCollection 2020. PMID 32265713
- [Background] Rasooli S, Moslemi F, Khaki A. Effect of Sub hypnotic Doses of Propofol and Midazolam for Nausea and Vomiting During Spinal Anesthesia for Cesarean Section. Anesth Pain Med. 2014 Sep 16;4(4):e19384. doi: 10.5812/aapm.19384. eCollection 2014 Oct. PMID 25346896
- [Background] Gouveia F, Oliveira C, Losa N. Acupuncture in the Management of Intraoperative Nausea and Vomiting. J Acupunct Meridian Stud. 2016 Dec;9(6):325-329. doi: 10.1016/j.jams.2016.09.005. Epub 2016 Sep 17. PMID 28010836
- [Background] Dewinter G, Staelens W, Veef E, Teunkens A, Van de Velde M, Rex S. Simplified algorithm for the prevention of postoperative nausea and vomiting: a before-and-after study. Br J Anaesth. 2018 Jan;120(1):156-163. doi: 10.1016/j.bja.2017.08.003. Epub 2017 Nov 23. PMID 29397124
- [Background] Shoar S, Esmaeili S, Safari S. Pain management after surgery: a brief review. Anesth Pain Med. 2012 Winter;1(3):184-6. doi: 10.5812/kowsar.22287523.3443. Epub 2012 Jan 1. PMID 24904790